CLINICAL TRIAL: NCT05001971
Title: Anlotinib Plus Penpulimab as Second-line Treatment for Patients With Small Cell Lung Cancer After Failure of Platinum-based Chemotherapy: a Single-arm, Multicenter Pilot Study
Brief Title: Anlotinib Plus Penpulimab as Second-line Treatment for Patients With Small Cell Lung Cancer After Failure of Platinum-based Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hunan Cancer Hospital (Other)
Collaborators: Fuzhou Pulmonary Hospital of Fujian (Other); Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTER-L041
Record Dates: First submitted 2021-01-29; First posted 2021-08-12 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — anlotinib; penpulimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib Plus Penpulimab (Experimental): Anlotinib (10mg qd po d1-14, 21 days per cycle) and Penpulimab (200mg ivgtt d1)
  Interventions: Drug: Anlotinib Plus Penpulimab

INTERVENTIONS:
Drug: Anlotinib Plus Penpulimab — Anlotinib: 10mg orally daily on day 1 to 14 of a 21-day cycle. Penpulimab: 200mg by intravenous drip on day 1 of a 21-day cycle.
  Other Names: Anlotinib & Penpulimab

SUMMARY:
Anlotinib is a multi-target receptor tyrosine kinase inhibitor in domestic research and development. It can inhibit the angiogenesis related kinase, such as VEGFR, FGFR, PDGFR, and tumor cell proliferation related kinase -c-Kit kinase. In the phase II ALTER1202 trial, patients who failed at least two kinds of systemic chemotherapy regimens (third line or beyond) or drug intolerance were treated with anlotinib or placebo, the anlotinib group PFS and OS were 4.1 months and 7.3 months, the placebo group PFS and OS were 0.7 months and 4.9 months. Therefore, the combination of Anlotinib and Penpulimab (a new PD-1 inhibitor) is attempted for the treatment of sensitive relapsed small-cell lung cancer patients who were failure in the first-line treatment of chemotherapy with platinum containing drugs, to further improve the patient's PFS or OS.

DETAILED DESCRIPTION:
This is a multicenter, single-arm, explorative clinical trial conducted in China to investigate the effectiveness and safety of Anlotinib Plus Penpulimab in patients with small cell lung cancer after failure of platinum-based chemotherapy.

Eligible patients will receive Anlotinib plus Penpulimab:

Anlotinib: 10mg orally daily on day 1 to 14 of a 21-day cycle. Penpulimab: 200mg by intravenous drip on day 1 of a 21-day cycle.

ELIGIBILITY:
Inclusion Criteria:

* signed and dated informed consent
* Small cell lung cancer pathologically confirmed, with measurable nidus (RECIST 1.1)
* have failed for first-line chemotherapy
* have a time interval ≥ 3 months between relapse and the end of the last systemic chemotherapy
* ECOG PS: 0-1, Expected Survival Time: Over 3 months
* main organs function is normal
* the woman patients of childbearing age who must agree to take contraceptive methods (e.g. intrauterine device, contraceptive pill or condom) during the research and within another 8 weeks after it; who are not in the lactation period and examined as negative in blood serum test or urine pregnancy test within 7 days before the research; The man patients who must agree to take contraceptive methods during the research and within another 8 weeks after it.

Exclusion Criteria:

* have used Anlotinib or other antiangiogenic drugs before
* have used Penpulimab or other anti-PD-1, anti-PD-L1, anti-CTLA-4 antibodies, as well as any other antibodies or drugs targeting T cell co-stimulatory or checkpoint pathways, such as ICOS or agonists (such as CD40, CD137, GITR, OX40, etc.)
* have failed for two times or beyond of platinum two drugs chemotherapy (except adjunctive chemotherapy, after which disease relapse or progression within 6 months，has been regarded as first-line therapy.)
* iconography (CT or MRI) shows obvious lung empty or necrotic tumor
* patients with brain or central nervous system metastases, including leptomeningeal disease, or CT/MRI examination revealed brain or leptomeningeal disease） (28 days before the random treatment has been completed and the symptoms of patients with brain metastases from stable can into the group, but need to the cerebral MRI, CT or vein angiography confirmed as without symptoms of cerebral hemorrhage)
* patients are participating in other clinical studies (other than non-interventional studies) less than 4 weeks from the end of the previous clinical study
* patients who had received chemotherapy, radiation, or other experimental anticancer therapy (except diphosphonate) within 4 weeks prior to the first dose of this study. Those who had previously received local radiotherapy were eligible if they met the following criteria: the end of radiotherapy was more than 4 weeks from the start of this study (brain radiotherapy was more than 2 weeks); In addition, the target lesions selected in this study were not in the radiotherapy area, or if the target lesion is within the radiotherapy area but progression has been confirmed
* other kinds of malignancies within 5 years or for now
* patients who have an active, known or suspected autoimmune disease, including a history of allogeneic organ transplantation, allogeneic hematopoietic stem cell transplantation, a history of being HIV positive, or a history of acquired immunodeficiency syndrome (AIDS)
* active or previously recorded inflammatory bowel disease (such as Crohn's disease, ulcerative colitis)
* have got non remissive toxic reactions derived from previous therapies, which is over level 1 in CTC AE (4.0), alopecia NOT included
* abnormal coagulation (INR > 1.5 or prothrombin time (PT) > ULN + 4 seconds or APTT ULN > 1.5), with bleeding tendency or be treated with thrombolysis and anticoagulation
* have clinical significant hemoptysis occurred within 3 months before enrollment (daily hemoptysis more than half tablespoonl; Or clinical significant bleeding symptoms or bleeding tendency in the 4 weeks prior to grouping, such as gastrointestinal bleeding, hemorrhagic gastric ulcer (including gastrointestinal perforation and/or fistula, but gastrointestinal perforation or fistula has been surgically removed, admission is allowed), baseline fecal occulted blood ++ or above, unhealed wounds, ulcers or fractures, etc
* urine routines show urine protein≥ ++, or urine protein quantity≥ 1.0 g during 24 hours
* uncontrollable hypertensive (SBP≥ 160 mmHg, DBP≥100 mmHg, despite the best drug treatment)
* patients with severe cardiovascular disease: grade II or above myocardial ischemia or myocardial infarction, poorly controlled arrhythmia; According to NYHA standard, grade III to IV cardiac insufficiency, or echocardiography indicates left ventricular ejection fraction (LVEF) < 50%;
* patients with NCI-CTCAE grade II or greater peripheral neuropathy, except due to trauma
* Interstitial lung disease, uncontrolled medium to large serosal effusion (including pleural effusion, ascites, and pericardial effusion) after pumping treatment, aggravated chronic obstructive pulmonary disease, active pulmonary infection and/or acute bacterial or fungal respiratory disease requiring intravenous antibiotic treatment within 28 days
* have an obvious factor influencing oral drug absorption, such as unable to swallow, chronic diarrhea and intestinal obstruction, etc
* have venous thromboembolism events within 6 months before enrollment, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism, etc
* have received live or attenuated vaccine within 30 days prior to the initial administration of Penpulimab, or was scheduled to receive live or attenuated vaccine during the study
* patients who have known a history of severe hypersensitivity to other monoclonal antibodies
* patients who have known a history of psychotropic substance abuse, alcohol abuse, or drug abuse
* uncontrolled active hepatitis after treatment (Hepatitis B: HBsAg positive and HBV DNA more than 1 x 10^4 copy /ml; Hepatitis C: HCV RNA is positive and liver function is abnormal); Combined with hepatitis b and hepatitis c infection
* serious diseases that endanger patients' safety or affect patients' completion of research, according to the researchers' judgment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2021-01-30 (Actual); Primary Completion 2025-01-21 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
ORR | up to 24 months
  Objective Response Rate

SECONDARY OUTCOMES:
PFS | each 42 days up to PD or death (up to 24 months)
  Progress free survival
OS | From randomization until death (up to 24 months)
  Overall Survival
DCR | each 42 days up to intolerance the toxicity or PD or death (up to 24 months)
  Disease Control Rate
Safety (Number of Participants with Adverse Events as a Measure of Safety and Tolerability） | Until 21 day safety follow-up visit
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Nong Yang, PhD, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Nong Yang, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion
Access Criteria: Data access requests will be reviewed by an external indepentent Review Panel. Requesdtors will be required to sign a Data Access Agreement.